CLINICAL TRIAL: NCT00799578
Title: A Preliminary Study to Evaluate Cysteamine Therapy in Human Subjects With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joel Lavine (Other)
Collaborators: Raptor Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor-Investigator, Joel Lavine, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-1699
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Fatty Liver
Keywords: NASH, NAFLD,nonalcoholic steatohepatitis
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cystagon-EC (Experimental)
  Interventions: Drug: Cysteamine

INTERVENTIONS:
Drug: Cysteamine — Drug is in enteric-coated capsule form. The dosage will begin at 1g/m-squared body surface area with a maximum dose of 1000mg twice daily. Treatment period is 3-6 months.

SUMMARY:
The purpose of this study is to determine whether cysteamine will effectively reduce or reverse the biologic markers of steatohepatitis in patients.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) steatohepatitis represents a spectrum of disease occurring in the absence of alcohol abuse. It is characterized by the presence of steatosis and may represent a hepatic manifestation of the metabolic syndrome (including obesity, diabetes and hypertriglyceridemia). NAFLD is linked to insulin resistance, it causes liver disease in adults and children and may ultimately lead to cirrhosis (Skelly et al., 2002). The histologic spectrum of NAFLD ranges from the relatively benign isolated predominantly macrovesicular steatosis (i.e., nonalcoholic fatty liver or NAFL) to steatohepatitis (NASH) (Angulo, & Lindor, 2002). The latter is characterized by the histologic presence of steatosis, cytological ballooning, scattered inflammation and pericellular fibrosis(Contos & Sanyal, 2002). Estimates of prevalence among children can be inferred from pediatric obesity data and the knowledge that 85% of children with NAFLD are obese. Data from the National Health and Nutrition Examination Survey has revealed a threefold rise in the prevalence of childhood and adolescent obesity over the past 35 years; data from 2000 suggests that 14-16% children between 6-19yrs age are obese with a BMI >95% (Fishbein, Miner, Mogren & Chalekson, 2003), and also the fact that 85% of children with NAFLD are obese.

Treatment of NASH currently revolves around the reduction of the two main pathogenetic factors, namely, fat accumulation within the liver and excessive accumulation of free radicals causing oxidative stress. Glutathione (gamma-glutamyl-cysteinyl-glycine; GSH) is a major endogenous antioxidant and its depletion is implicated in the development of hepatocellular injury (Wu, Fang, Yang, Lupton & Turner, 2004). Glutathione itself is does not enter easily into cells, even when given in large amounts. However, glutathione precursors do enter into cells and have been shown to be effective in the treatment of conditions such as acetaminophen toxicity by preventing significant GSH depletion (Prescott & Critchley, 1983). Examples of GSH precursors include cysteine, N-acetylcysteine, methionine and other sulphur-containing compounds such as cysteamine (Prescott, Park & Proudfoot, 1976). Studies have demonstrated that orally and intravenously administered cysteamine in mice and humans is effective in acetaminophen-induced hepatocellular injury (Prescott, 1972; Prescott, Stewart & Proudfoot, 1978; Mitchell, Thorgeirsson, Potter, Jollow & Keiser, 1974). Another study where N-acetylcysteine was used to treat NASH over a period of 4-12 weeks demonstrated improved amniotransferase levels (Pamuk & Sonsuz, 2003), suggesting that increasing GSH levels may have a hepato-protective role and may be useful in the treatment of NASH. A possible mode of action of cysteamine is that it might react with extracellular cystine to form cysteine which then is readily taken up into the cell and transformed into GSH.

Recent studies have suggested that the essential amino acid cysteine is a major limiting factor for GSH synthesis and that factors (e.g., insulin and growth factors) that stimulate cysteine uptake by cells generally result in increased intracellular GSH levels (Lyons et al., 2000; Lu, 2000).

Cysteamine, a GSH precursor, is currently available and is used in the treatment of cystinosis, an intra-lysosomalcystine storage disorder. In cystinosis, cysteamine acts by converting cystine to cysteine and cysteine-cysteamine mixed disulfide which are the both able to leave the lysosome through the cysteine and lysine porters respectively (Gahl, Theone & Shneider, 2002). Within the cytosol the mixed disulfide can be reduced by its reaction with glutathione and the cysteine released can be used for further GSH synthesis. The synthesis of GSH from cysteine is catalyzed by two enzymes, gamma-glutamylcysteine synthetase and GSH synthetase. This pathway occurs in almost all cell types, with the liver being the major producer and exporter or GSH. The reduced cysteine-cysteamine mixed disulfide will also release cysteamine, which, in theory is then able to re-enter the lysosome, bind more cystine and repeat the process (Dohil et al., 2006). In a recent study in children with cystinosis, enteral administration of cysteamine resulted in increased plasma cysteamine levels, which subsequently caused prolonged efficacy in the lowering of leukocyte cystine levels (Dohil et al., 2006). This may have been due to "re-cycling" of cysteamine when adequate amounts of drug reached the lysosome. If cysteamine does act in this fashion, then GSH production may also be significantly enhanced.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed diagnosis of non-alcoholic steatohepatitis (within past 12 months)
* Ages 10 yrs and older
* Must swallow tablets on a regular basis
* ALT level >60 iu/L

Exclusion Criteria:

* Subjects with known hypersensitivity to cysteamine
* History, currently or within the past 3 months, of the following conditions:
* Pancreatitis
* Inflammatory bowel disease
* Malabsorption
* Unstable heart disease, e.g., myocardial infarction, heart failure, arrhythmias.
* Unstable diabetes mellitus
* Any bleeding disorder.
* Zollinger-Ellison syndrome
* Malignant disease
* Subjects whom maybe pregnant or have health issues that make it unsafe for them participate, or whose concomitant medical problems preclude them from committing to the study schedule.
* No specific NASH medical therapy for 3 months such as vitamin E, s-adenosyl methionine or metformin or other NAFLD study drugs.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego School of Medicine General Clinic Research Center, San Diego, California, United States

REFERENCES:
- [Background] Skelly AH, Arcury TA, Gesler WM, Cravey AJ, Dougherty MC, Washburn SA, Nash S. Sociospatial knowledge networks: appraising community as place. Res Nurs Health. 2002 Apr;25(2):159-70. doi: 10.1002/nur.10024. PMID 11933009
- [Background] Angulo P, Lindor KD. Non-alcoholic fatty liver disease. J Gastroenterol Hepatol. 2002 Feb;17 Suppl:S186-90. doi: 10.1046/j.1440-1746.17.s1.10.x. PMID 12000605
- [Background] Contos MJ, Sanyal AJ. The clinicopathologic spectrum and management of nonalcoholic fatty liver disease. Adv Anat Pathol. 2002 Jan;9(1):37-51. doi: 10.1097/00125480-200201000-00005. PMID 11756758
- [Background] Fishbein MH, Miner M, Mogren C, Chalekson J. The spectrum of fatty liver in obese children and the relationship of serum aminotransferases to severity of steatosis. J Pediatr Gastroenterol Nutr. 2003 Jan;36(1):54-61. doi: 10.1097/00005176-200301000-00012. PMID 12499997
- [Background] Wu G, Fang YZ, Yang S, Lupton JR, Turner ND. Glutathione metabolism and its implications for health. J Nutr. 2004 Mar;134(3):489-92. doi: 10.1093/jn/134.3.489. PMID 14988435
- [Background] Prescott LF, Critchley JA. The treatment of acetaminophen poisoning. Annu Rev Pharmacol Toxicol. 1983;23:87-101. doi: 10.1146/annurev.pa.23.040183.000511. PMID 6347057
- [Background] Prescott LF, Park J, Proudfoot AT. Cysteamine, L-methionine and D-penicillamine in paracetamol poisoning. J Int Med Res. 1976;4(4 Suppl):112-7. doi: 10.1177/14732300760040S420. No abstract available. PMID 1026552
- [Background] Prescott LF. Haemodialysis in paracetomol self-poisoning. Lancet. 1972 Sep 23;2(7778):652. doi: 10.1016/s0140-6736(72)93038-3. No abstract available. PMID 4116795
- [Background] Prescott LF, Stewart MJ, Proudfoot AT. Cysteamine or N-acetylcysteine for paracetamol poisoning? Br Med J. 1978 Apr 1;1(6116):856-7. doi: 10.1136/bmj.1.6116.856-a. No abstract available. PMID 638489
- [Background] Mitchell JR, Thorgeirsson SS, Potter WZ, Jollow DJ, Keiser H. Acetaminophen-induced hepatic injury: protective role of glutathione in man and rationale for therapy. Clin Pharmacol Ther. 1974 Oct;16(4):676-84. doi: 10.1002/cpt1974164676. No abstract available. PMID 4417718
- [Background] Lyons J, Rauh-Pfeiffer A, Yu YM, Lu XM, Zurakowski D, Tompkins RG, Ajami AM, Young VR, Castillo L. Blood glutathione synthesis rates in healthy adults receiving a sulfur amino acid-free diet. Proc Natl Acad Sci U S A. 2000 May 9;97(10):5071-6. doi: 10.1073/pnas.090083297. PMID 10792033
- [Background] Lu SC. Regulation of glutathione synthesis. Curr Top Cell Regul. 2000;36:95-116. doi: 10.1016/s0070-2137(01)80004-2. No abstract available. PMID 10842748
- [Background] Gahl WA, Thoene JG, Schneider JA. Cystinosis. N Engl J Med. 2002 Jul 11;347(2):111-21. doi: 10.1056/NEJMra020552. No abstract available. PMID 12110740
- [Background] Dohil R, Fidler M, Barshop BA, Gangoiti J, Deutsch R, Martin M, Schneider JA. Understanding intestinal cysteamine bitartrate absorption. J Pediatr. 2006 Jun;148(6):764-9. doi: 10.1016/j.jpeds.2006.01.050. PMID 16769383
- [Background] Pamuk GE, Sonsuz A. N-acetylcysteine in the treatment of non-alcoholic steatohepatitis. J Gastroenterol Hepatol. 2003 Oct;18(10):1220-1. doi: 10.1046/j.1440-1746.2003.03156.x. No abstract available. PMID 12974918
- [Derived] Dohil R, Schmeltzer S, Cabrera BL, Wang T, Durelle J, Duke KB, Schwimmer JB, Lavine JE. Enteric-coated cysteamine for the treatment of paediatric non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2011 May;33(9):1036-44. doi: 10.1111/j.1365-2036.2011.04626.x. Epub 2011 Mar 13. PMID 21395631
- See also: Related Info — http://www2.niddk.nih.gov/
- See also: Related Info — http://win.niddk.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Biopsy proven children with nonalcoholic fatty liver disease from fatty liver clinic at University of California, San Diego
Pre-assignment Details: Not on other therapy for NAFLD
Period: Overall Study
Arm/Group | Cystagon-EC
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cystagon-EC
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Normalization or >50% of Serum ALT Levels From Baseline
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Number of Improved Subjects
Number analyzed (Participants) | 11
participants | 7

ADVERSE EVENTS:
Arm/Group | Number of Improved Subjects
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No